CLINICAL TRIAL: NCT06878651
Title: Investigation of the Immediate Effects of Whole Body Vibration Training on Balance, Dual Task and Gait in Individuals with Diabetic Neuropathy
Brief Title: The Instant Effect of Whole Body Vibration in Diabetics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Gulhane Training and Research Hospital (Other Government); Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-553
Record Dates: First submitted 2025-02-21; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetus Mellitus; Diabetic Foot Ulcer; Diabetic Neuropathic Ulcer
Keywords: Diabetic Foot; Diabetes Mellitus; Foot Ulceration; Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: This study follows an interventional pre-post experimental design, focusing on the immediate effects of whole-body vibration (WBV) on balance, gait, and dual-task performance in patients with diabetic foot. The interventional model used is a single-group pretest-posttest design, where participants undergo a single WBV session, and their performance metrics are assessed before and after the intervention.
Masking Description: In this study, no formal masking (blinding) is applied, as the nature of the intervention (whole-body vibration) makes it challenging to conceal from participants and assessors. However, alternative approaches to minimizing bias are considered.
  Masking in the Study Participants: Not masked. Since WBV is a physical intervention, participants are aware they are receiving treatment, making blinding impossible.
  Researchers Conducting the Intervention: Not masked. The investigators administering WBV are aware of the intervention settings and participant exposure.
  Outcome Assessors (If Different from Researchers): Not masked. The same researchers conducting the intervention may also conduct pre- and post-tests, increasing the potential for observer bias.
  Data Analysts: Potential for masking. If feasible, data analysis could be conducted by an independent researcher blinded to the intervention phase (pre- or post-WBV) to reduce bias in interpreting results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): In the Control Group, balance assessment with the Timed Up and Go Test, evaluation of dual task performance with the Dual Task Cost Gap Formula, and gait assessment with the 1 Minute Walk Test will be performed.
- Whole Body Vibration Training Group (Experimental): For the Whole Body Vibration Training Group, balance, dual task performance and gait will be evaluated. These participants will be evaluated before and after 10 minutes of vibration application.
  Interventions: Device: The Whole Body Vibration

INTERVENTIONS:
Device: The Whole Body Vibration — Whole Body Vibration device may positively affect balance, dual-tasking and gait parameters by increasing the sensory input received under the sole in individuals diagnosed with diabetic foot. In individuals diagnosed with diabetic foot, the sensory/vibration perception threshold of individuals decreases due to the disease, so the balance of individuals is impaired. This may cause these individuals to experience gait disturbances in daily life. There are almost no studies in the literature on the use of whole body vibration for this patient group. This study will discuss the applicability of whole body vibration in the clinic for individuals diagnosed with diabetic foot and that it can be an additional adjunct to treatment.
  Arms: Whole Body Vibration Training Group

SUMMARY:
Overview of Diabetes and Its Complications:

* Diabetes is a chronic health issue that can lead to various complications, affecting human health negatively. One of these complications is diabetic peripheral neuropathy (DPN), which results from hyperglycemia and affects peripheral nerves. This can lead to sensory loss, motor dysfunction, and ultimately, disability.
* The complications from diabetes can result in the loss of function and disability, affecting various systems, including the nervous system (e.g., retinopathy, neuropathy, and atherosclerosis).

Peripheral Neuropathy in Diabetes:

* DPN occurs due to damage to peripheral nerves caused by hyperglycemia. Over time, it affects the small unmyelinated fibers responsible for pain and temperature sensations, leading to axonal degeneration and demyelination, causing sensory loss.
* In later stages, motor dysfunction can also occur, impacting intrinsic foot muscles, leading to muscle weakness and atrophy.

Whole Body Vibration (WBV) Therapy:

* WBV is a therapeutic method that uses mechanical vibrations from a vibrating platform to stimulate muscle contractions. It is being researched for its effects on managing diabetic neuropathy and related complications.
* Studies have shown that WBV can improve balance, functional independence, and postural stability in patients with diabetes, potentially serving as an alternative or complement to traditional balance exercises.
* A randomized controlled trial compared the effects of WBV and Tai Chi on postural balance and found that WBV was more effective in promoting functional independence and balance.

Impact on Sensory Function and Balance:

* As DPN progresses, sensory loss may prevent patients from noticing injuries, which could lead to severe complications. A study conducted in 2017 showed that WBV improved vibration perception thresholds (VPT) in patients with type 2 diabetes and peripheral neuropathy, indicating improved sensory function, which is crucial for maintaining balance and walking.
* This improvement is thought to be linked to increased blood circulation in peripheral tissues and improved glucose levels due to WBV therapy.

Dual Task Performance and WBV:

- Dual-task performance, which involves performing cognitive and motor tasks simultaneously, is typically impaired in patients with diabetic neuropathy, leading to difficulties in daily activities. WBV has shown potential in improving muscle strength and balance, which could enhance patients' ability to perform dual tasks more effectively.

Research Findings:

* Several studies have demonstrated that WBV training can significantly improve both static and dynamic balance in patients with diabetic neuropathy. Given that balance issues are common in these patients and contribute to a higher risk of falls, these improvements are particularly important.
* The literature emphasizes the need for continued research to clarify the physiological mechanisms behind WBV's effects on sensory feedback mechanisms, which are essential for postural control.

Need for Further Research:

* Despite promising findings, some studies have pointed out the need for more research to validate the clinical efficacy of WBV for managing chronic complications like neuropathic pain and improving quality of life in diabetic patients.
* There is a need for better-designed studies to confirm the long-term benefits of WBV training in diabetic patients and to develop standardized protocols for its use.

Proposed Study:

* A planned study aims to investigate the immediate effects of WBV on balance, dual-task performance, and walking in individuals with type 2 diabetes and peripheral neuropathy. The study will include 40 patients who meet specific inclusion criteria, with participants randomized into two groups (WBV training group and control group).
* Data will be collected on participants' balance performance (using the Timed Up and Go test), dual-task performance (using a dual-task cost formula), and walking features (using the 1-minute walk test). The results will be analyzed using SPSS software.

Methodology:

- The study will use random assignment and include a control group to evaluate the immediate effects of WBV. Data collection will include assessments of balance, dual-task performance, and walking capabilities before and after WBV treatment.

DETAILED DESCRIPTION:
Sure! Here's a more detailed and extended version of the summary:

Diabetes is a chronic health condition that can lead to various complications, affecting many aspects of human health. One of the significant complications resulting from diabetes is peripheral neuropathy, which is caused by hyperglycemia-induced damage to peripheral nerves. Over time, this condition results in axonal degeneration and demyelination, particularly affecting small unmyelinated fibers responsible for pain and temperature sensation, leading to sensory loss. In advanced stages, it can result in motor dysfunction, which particularly affects intrinsic foot muscles, leading to muscle weakness and atrophy. Peripheral neuropathy can significantly impair balance, dual-task performance, and gait, all of which are crucial for maintaining functional independence and mobility in diabetic patients.

The effect of Whole Body Vibration (WBV) training on these aspects has been an emerging research area. WBV, which uses mechanical vibrations produced by a vibrating platform to stimulate muscle contractions, has shown potential benefits in improving balance, dual-task performance, and gait in individuals with diabetic neuropathy. Several studies have suggested that WBV can serve as a complementary or superior alternative to traditional balance training exercises. For instance, a randomized controlled trial comparing WBV and Tai Chi in diabetic patients found that WBV was more effective than Tai Chi in promoting functional independence and improving balance.

In patients with diabetic peripheral neuropathy (DPN), sensory loss may prevent them from recognizing injuries, leading to severe complications. A study from 2017 explored the impact of WBV on vibration perception thresholds (VPT) in patients with type 2 diabetes and peripheral neuropathy, finding significant improvements in VPT, which indicated enhanced sensory function, critical for maintaining balance and gait. This improvement was attributed to increased blood circulation in peripheral tissues and better glucose control, which positively influenced sensory feedback mechanisms crucial for postural control.

Moreover, WBV has been shown to improve both static and dynamic balance in individuals with DPN, which is vital for reducing fall risks in these patients. The improvements in balance are believed to result from muscle contraction stimulation and the proprioceptive feedback provided by the vibrations. Furthermore, dual-task performance, which is often impaired in patients with DPN due to the difficulty of performing cognitive and motor tasks simultaneously, might also improve with WBV. This improvement could help patients perform better in daily activities that require multitasking, such as walking while engaging in cognitive tasks.

In the existing literature, there is evidence that WBV training enhances balance and walking ability in diabetic patients, although there is a gap in research that simultaneously addresses balance, dual-task performance, and gait parameters in type 2 diabetes patients. A systematic review conducted by Robinson and colleagues in 2018 noted the potential benefits of WBV in managing neuropathic pain and improving the quality of life for DPN patients, although the clinical effectiveness of WBV as an intervention for DPN remains unclear. This highlights the need for further research to clarify the therapeutic role of WBV in this patient population.

The growing body of evidence supporting the effectiveness of WBV in improving balance, dual-task performance, and gait in diabetic neuropathy patients suggests that it could be a promising therapeutic approach. The literature emphasizes the necessity for continued research to establish standardized protocols and further explore the physiological mechanisms underlying the potential benefits of WBV in this sensitive population. More well-designed studies are needed to confirm the long-term benefits of WBV training and validate its role in the management of diabetic neuropathy. By incorporating WBV into treatment programs, physiotherapists can provide a more holistic approach to managing diabetic neuropathy, enhancing functional outcomes and potentially improving the quality of life for affected individuals.

This study aims to provide a comprehensive overview of the immediate effects of WBV on balance, dual-task performance, and gait in individuals with diabetic neuropathy. The research will be conducted as a single-blind randomized controlled trial involving 40 participants diagnosed with diabetic peripheral neuropathy, all of whom will be selected voluntarily from a specialized diabetes foot clinic. Participants will be randomly assigned to either the experimental group (receiving WBV training) or the control group, with baseline and post-intervention assessments conducted to measure changes in balance, dual-task performance, and gait. Various tools, including the Timed Up and Go test, the Dual Task Costs formula, and the 1-minute walk test, will be used to assess these parameters. The study will utilize appropriate statistical analyses, including comparisons within and between groups, and will follow ethical guidelines, ensuring informed consent from all participants.

By evaluating these parameters, the study aims to contribute to the understanding of how WBV can improve functional outcomes in individuals with diabetic neuropathy and guide future therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients aged 40-75 years,
* Having a score of 13-29 on the Michigan Questionnaire (intermediate level),
* Having a Mini Mental Test score of 24 and above,
* Having an HbA1C <8.5%, having controlled blood glucose levels in the last three months,
* Being able to walk independently
* Volunteering to participate in the study.

Exclusion Criteria:

* Those with diabetic infected wounds,
* Those with neurological diseases other than diabetic neuropathy,
* Those with rheumatoid arthritis, vestibular system disorders, visual
* Impairments, those with a history of trauma, injury and surgery,
* Those with knee or hip replacement,
* Those with a history of epilepsy and cognitive problems.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Balance Performance | For the control group the test will be administered once at baseline and 10 minute later on the same day . In the vibration training group, it will be administered at Baseline (Before WBV) and Immediately After WBV (within 5 minutes).
  Change in balance performance assessed using the Timed Up and Go (TUG) test. The test measures the time taken (in seconds) to rise from a chair, walk 3 meters, turn, and return to sit. Lower times indicate better balance and functional mobility.
Gait Performance | For the control group (one-time assessment at baseline and 10 minutes later), For the WBV Training Group Baseline (Pre-WBV) and Immediately Post-WBV
  Change in walking capacity measured by the 1-Minute Walk Test. Total distance walked (in meters) is recorded, with greater distances indicating better walking endurance and gait function.

SECONDARY OUTCOMES:
Functional Mobility (Timed Up and Go Test - TUG) | Start (Before WBV) and Immediately After WBV (within 10 minutes)
  Change in functional mobility and dynamic balance measured by the Timed Up and Go (TUG) test. The outcome is the time taken (in seconds) to complete the test. A shorter time after WBV indicates improved mobility and balance.
Cognitive-Motor Performance (Dual-Task Timed Up and Go Test - DT-TUG) | Start (Before WBV) and Immediately After WBV (within 5 minutes)
  Change in cognitive-motor performance measured by the Dual-Task Timed Up and Go (DT-TUG) test. Performance is evaluated through the dual-task gap formula, reflecting the percentage increase in TUG time during the cognitive task. A reduced dual-task gap post-WBV suggests better cognitive-motor integration.
Walking Capacity (1-Minute Walk Test) | Start (Before WBV) and Immediately After WBV (within 5 minutes)
  Change in walking distance measured by the 1-Minute Walk Test. The total distance walked (in meters) reflects gait capacity, endurance, and speed. An increased distance after WBV indicates enhanced walking performance.

OTHER OUTCOMES:
Patient Demographics and Clinical Characteristics | In the study group, the whole body vibration device will be applied by vibrating under the floor at baseline and after 10 minutes in the same day.
  Other pre-specified outcomes include patient demographics and clinical characteristics, such as age, weight, gender, duration of diabetes diagnosis, and insulin use, to explore their potential influence on functional outcomes. Glycemic control markers, including the most recent blood glucose value and HbA1c percentage, will be recorded to assess metabolic status. Cognitive function will be evaluated using the Mini-Mental State Examination (MMSE), while peripheral neuropathy severity will be determined through the Michigan Neuropathy Screening Instrument (MNSI) and clinical staging of diabetic neuropathy. Additionally, the use of assistive devices, such as walking aids or orthotics, will be noted, as these factors may influence balance, gait, and dual-task performance. Collectively, these measures provide a comprehensive clinical context to better understand the factors that may modulate the effects of whole-body vibration therapy.
Dual-Task Performance | For the control group the test will be administered baseline and 15 minutes later in the same day. In the vibration training group, it will be administered at Baseline (Before WBV) and Immediately After WBV (within 5 minutes).
  Change in cognitive-motor function measured using the Dual-Task Timed Up and Go (DT-TUG) test. The dual-task gap formula is applied to calculate the percentage difference between single-task and dual-task states, reflecting the cognitive load's impact on mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Şahan, Study Director — Gülhane Sağlık Bilimleri Üniversitesi; Dilek N Kara, Principal Investigator — Bağlı Olmayan; Kerim B Profesör Doktor, Study Chair — Gulhane Training and Research Hospital
Locations (1):
- Gülhane Eğitim ve Araştırma Hastanesi, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is a clause in our consent form about the use of the information for other studies. This is something that is emphasized by our university. Therefore, in order to protect patient rights, it is not possible to share information without patient consent.

REFERENCES:
- [Background] Sohrabzadeh E, Kalantari KK, Naimi SS, Daryabor A, Akbari NJ. The immediate effect of a single whole-body vibration session on balance, skin sensation, and pain in patients with type 2 diabetic neuropathy. J Diabetes Metab Disord. 2021 Nov 25;21(1):43-49. doi: 10.1007/s40200-021-00933-w. eCollection 2022 Jun. PMID 35673453
- [Background] Jamal A, Ahmad I, Ahamed N, Azharuddin M, Alam F, Hussain ME. Whole body vibration showed beneficial effect on pain, balance measures and quality of life in painful diabetic peripheral neuropathy: a randomized controlled trial. J Diabetes Metab Disord. 2019 Dec 21;19(1):61-69. doi: 10.1007/s40200-019-00476-1. eCollection 2020 Jun. PMID 32550157